CLINICAL TRIAL: NCT03529656
Title: The Safety and Efficacy of Early Rehabilitation Program in Immediate Liver Transplant Patients
Brief Title: The Early Rehabilitation Program in Post-LT Pts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, Associate professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AsanMC-LT rehab
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: ICU-acquired Weakness
Keywords: Liver transplantation; rehabilitation; ICU acquired weakness
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-ERP (No Intervention): A group of patients who underwent liver transplantation surgery before the early rehabilitation program
- Post-ERP (Experimental): A group of immediate liver transplant patients who had an early rehabilitation program in ICU care
  Interventions: Behavioral: Early rehabilitation program for liver transplantation

INTERVENTIONS:
Behavioral: Early rehabilitation program for liver transplantation — Deliver the one of 5-step early rehabilitation program for immediate liver transplant pts on weekday
  Arms: Post-ERP

SUMMARY:
The purpose of this study is to determine whether an early rehabilitation program for immediate liver transplant patients is safe and effective in preventing critical care illness and intensive care unit acquired weakness.

DETAILED DESCRIPTION:
Patients with liver transplantation (LT) have poor general condition before surgery and require ICU care for a certain period. For those patients, the side effects of ICU care such as intensive care unit-acquired weakness (ICU-AW), critical illness polyneuropathy (CIP) are well known. Therefore, we access the safety and efficacy of early rehabilitation program (ERP) in liver transplant recipients.

Patients were retrospectively selected for the Pre-ERP group (2014.05-2014.10) and for the Post-ERP group (2015.10-2016.03). During the period of 6 months, 136 patients and 100 patients underwent LT, and 65, 62 patients were enrolled after exclusion. Forty patients from the each group were compared after propensity score matching (PSM).

ELIGIBILITY:
Inclusion Criteria:

* immediate post liver transplant patients

Exclusion Criteria:

* patients who transferred to sub-ICU within 72 hours re-liver transplantation case wound, mental problem post op bleeding unstable vital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
ICU day (days) | up to 60 days
ventilator day (days) | up to 60 days

SECONDARY OUTCOMES:
Time to start rehabilitation from ICU admission (days) | up to 2 weeks
in-hospital LOS (days) | up to 24 weeks
hospital readmission rate after surgery (%) | 1 year follow up from the surgery
1 year mortality rate (%) | 1 year follow up from the surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cortazzo MH, Helkowski W, Pippin B, Boninger ML, Zafonte R. Acute inpatient rehabilitation of 55 patients after liver transplantation. Am J Phys Med Rehabil. 2005 Nov;84(11):880-4. doi: 10.1097/01.phm.0000184093.53032.ed. PMID 16244526
- [Result] Kothari AN, Yau RM, Blackwell RH, Schaidle-Blackburn C, Markossian T, Zapf MA, Lu AD, Kuo PC. Inpatient Rehabilitation after Liver Transplantation Decreases Risk and Severity of 30-Day Readmissions. J Am Coll Surg. 2016 Jul;223(1):164-171.e2. doi: 10.1016/j.jamcollsurg.2016.01.061. Epub 2016 Feb 13. PMID 27049779
- [Result] Maffei P, Wiramus S, Bensoussan L, Bienvenu L, Haddad E, Morange S, Fathallah M, Hardwigsen J, Viton JM, Le Treut YP, Albanese J, Gregoire E. Intensive Early Rehabilitation in the Intensive Care Unit for Liver Transplant Recipients: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1518-1525. doi: 10.1016/j.apmr.2017.01.028. Epub 2017 Mar 6. PMID 28279659